CLINICAL TRIAL: NCT01187095
Title: A Randomized Controlled Intervention Study: The Effect of Expressive Writing on Psychosocial Stress and Pregnancy Results With Couples Undergoing In Vitro Fertility(IVF) Treatment Due to Involuntary Childlessness.
Brief Title: Involuntary Childlessness and Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Yoon Frederiksen, PhD.-fellowship, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EWI-2008-41-1869
Record Dates: First submitted 2010-07-09; First posted 2010-08-23 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Infertility
Keywords: Involuntary childlessness; Infertility; IVF; EWI; Couples in IVF treatment; Psychosocial intervention
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- counselling (Experimental): Does couples in IVF treatment benefit from emotional disclosure
  Interventions: Behavioral: Expressive writing
- Control (Active Comparator): Neutral writing exercise
  Interventions: Behavioral: Active ctrl

INTERVENTIONS:
Behavioral: Expressive writing — 3 consecutive days of writing
  Other Names: EWI
  Arms: counselling
Behavioral: Active ctrl — Control
  Arms: Control

SUMMARY:
Many couples experience involuntary childlessness and seek treatment at fertility clinics. Going through treatment procedures can be very challenging, time consuming and emotionally demanding.

Psychosocial intervention might have a soothing and healing effect on both behavior as well on physical matters. Hence, the investigators would like to investigate whether Expressive Writing Intervention (EWI) has an effect on stress management as well as on the pregnancy rate for couples who are going through fertility treatment.

DETAILED DESCRIPTION:
Background:

Around 10-14 % of all couples are experiencing involuntary childlessness. Most of these couples will be referred to the public health clinics in order to receive help by means of fertility treatment e.g. in vitro fertility (IVF) and numbers from the National board of Health indicates that the number is rising. It is well known that involuntary childlessness pose an enduring psychosocial burden and strain with feelings of hopelessness, despair, anger and frustration as well as anxiety and sadness. Much research points out that couples that receive IVF treatment to a great extent often experience stress and strong emotional oscillations during the treatment procedures. Some studies indicate that negative feelings as described above might have a negative impact on the chances of becoming pregnant. In spite of these findings there are only conducted very few controlled studies of intervention with this patient group, which might explain why it is still unclear whether infertile couples can benefit from therapeutic intervention.

A growing number of studies in the area of health psychology has suggested that interventions where the participants has the opportunity to express themselves in writing about feelings, so-called Expressive Writing Intervention (EWI) seem to have a positive effect on physical health as well as mental well-being.

Methods:

Couples starting with their IVF treatment at the Fertility Clinic, Skejby Hospital will be invited to participate in the research project. Approximately 400 couples are expected to begin treatment during a one year period (We would like to enrol at least 144 couples). They will be randomized into a EWI group (writing about fertility related topics - emotional disclosure) and a control group (writing about neutral topics non-emotional disclosure).

Inclusion criteria:

* Heterosexual couples as well as Homosexual couples
* 1st, 2nd and 3rd treatment cycles
* Can read and understand Danish
* Aged 18-40 years

Exclusion criteria:

• Patients with genetic diseases (PGD patients)

The investigators would like to know more about whether EWI has an effect on:

1. The extent of psychosocial strain - does change happen in life satisfaction, emotional state and reactions, as well as with thoughts about childlessness and treatment.
2. The result of the IVF treatment (pregnancy/non pregnancy)
3. The adaptation to the (negative) treatment outcome - the impact of having participated in an EWI intervention group.

Furthermore mediators and moderators will be explored.

ELIGIBILITY:
Inclusion Criteria:

* heterosexual couples lesbian couples

Exclusion Criteria:

* couples; where one of them suffers from a genetic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 298 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Zachariae, prof.med.,, Principal Investigator — University of Aarhus
Locations (1):
- Department of Psychology, Aarhus University, Aarhus, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philipsen MT, Knudsen UB, Zachariae R, Ingerslev HJ, Hvidt JEM, Frederiksen Y. Sleep, psychological distress, and clinical pregnancy outcome in women and their partners undergoing in vitro or intracytoplasmic sperm injection fertility treatment. Sleep Health. 2022 Apr;8(2):242-248. doi: 10.1016/j.sleh.2021.10.011. Epub 2021 Dec 20. PMID 34949542
- [Derived] Frederiksen Y, O'Toole MS, Mehlsen MY, Hauge B, Elbaek HO, Zachariae R, Ingerslev HJ. The effect of expressive writing intervention for infertile couples: a randomized controlled trial. Hum Reprod. 2017 Feb;32(2):391-402. doi: 10.1093/humrep/dew320. Epub 2016 Dec 21. PMID 28007790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Couples were recruited from November 2010 through July 2012. Recruitment took place at the following three Danish fertility clinics: The Fertility Clinic at Aarhus University Hospital, Skive Fertility Clinic, Skive; Brædstrup Fertility Clinic, Brædstrup.
Groups:
- Counselling: Do couples in IVF treatment benefit from emotional disclosure
  Expressive writing: 3 consecutive days of writing
Period: Overall Study
Arm/Group | Counselling | Control
Started | 153 | 142
Completed | 108 | 108
Not Completed | 45 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counselling | Control | Total
Number analyzed (Participants) | 153 | 142 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The rows indicate the age dependent on gender
  years
    Women: number analyzed (Participants) | 83 | 80 | 163
    Women | 31.9 (4.4) | 32.9 (4.8) | 32.3 (4.5)
    Partners: number analyzed (Participants) | 70 | 62 | 132
    Partners | 33.9 (5.9) | 34.7 (6.2) | 34.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported data
  Participants
    Female | 83 | 80 | 163
    Male | 70 | 62 | 132
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 153 | 142 | 295

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Expressive Writing Intervention on Fertility Related Stress
Description: The COMPI 14-item self-rating instrument has been developed to capture specific thoughts and feelings in relation to involuntarily childlessness, which may lead to distress on 4-point and 5-point Likert scales. Responses cover personal, social, and marital domains with total scores ranging between 14 - 38, and higher scores indicating higher levels of infertility-related distress. Internal consistency (Cronbach's alpha) in the present study was 0.89 and the baseline to post-intervention test-retest correlation was 0.84. For the sub-domains the reliability of the scales were as follows; personal domain α=0.86, social domain α=0.83 and marital domain α=0.73.
Time Frame: follow-up 2 (3 months)
Population: Couples undergoing IVF or ICSI fertility treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counselling | Control
Number analyzed (Participants) | 153 | 142
units on a scale
  Baseline | 17.2 (9.0) | 15.7 (9.1)
  Follow up 1 | 17.4 (10.2) | 17.1 (9.8)
  Follow up 2 | 18.7 (9.5) | 17.6 (10.1)
Statistical Analysis 1: Comparison: Counselling vs Control; Test type: Non-Inferiority or Equivalence — Estimation parameter; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Counselling vs Control; Test type: Superiority; p < 0.05, Regression, Logistic

2. Secondary Outcome: Pregnancy Rate
Description: How many women achieved pregnancy in each arm
Time Frame: measured at follow-up (t3) 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Counselling | Control
Number analyzed (Participants) | 83 | 80
Participants | 42 | 39

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Counselling | Control
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes